CLINICAL TRIAL: NCT00605319
Title: An Open Label Study to Measure the Efficacy of Fesoterodine (Toviaz) on Continued Detrusor Overactivity in Patients That Have Undergone Treatment for Bladder Outlet Obstruction
Brief Title: An Open Label Study to Measure Efficacy of Fesoterodine (Toviaz) Post Surgery for Benign Prostatic Hyperplasia
Acronym: Toviaz
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0506007934; 2005-0202
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Bladder Outlet Obstruction
Keywords: BPH; BOO
MeSH Terms: conditions — Urinary Bladder Neck Obstruction | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toviaz (Fesoterodine) (Other): Toviaz 4mg to 8mg
  Interventions: Drug: Toviaz (Fesoterodine)

INTERVENTIONS:
Drug: Toviaz (Fesoterodine) — 4mg to 8mg by mouth once daily
  Other Names: Toviaz

SUMMARY:
The subjects who have symptoms of overactive bladder (many trips to the bathroom, and urgency with or without the inability to hold your urine until you get to the toilet) are invited to participate in this research study.

DETAILED DESCRIPTION:
Overactive bladder is a common sequelae of long-term bladder outlet obstruction in men. Unfortunately, it does not often resolve after treatment of the obstruction (transurethral resection of the prostate). These patients are usually started empirically on alpha-blockers or occasionally anticholinergic agents, former used to treat enlarged prostate medically, and latter, to treat overactive bladder. We hypothesize that these patients would be significantly improved with a long-acting anticholinergic agent such as long acting Fesoterodine or Toviaz.

Earlier studies have shown that anticholinergic drugs seem to have a beneficial effect on symptoms of patients with bladder outlet obstruction and overactive bladder. In addition, anticholinergic drug Toviaz is not associated with increased incidence of complication like acute urinary retention, a state where patient is unable to empty the bladder as an adverse effect of the drug.

A large proportion of our patients that are undergoing treatment for bladder outlet obstruction also have overactive bladder. We propose an open label trial to evaluate the efficacy of Toviaz (fesoterodine) 4mg to 8 mg in patients that have continued symptoms of overactive bladder one month following transurethral resection of the prostate. Toviaz is an antimuscarinic and anticholinergic agent, and is a newer formulation of Detrol. Patients with overactive bladder on urodynamic test preoperatively will be considered. If these patients continue to have symptoms at the one-month post-operative visit, they will be enrolled into the study. We expect a total of 25 patients to be enrolled within 4 months. All patients will receive Toviaz 4mg to 8 mg. The patients will be followed at 3 months post-op, 4 months post-op, and 7 months post-op. At each post-op visit, the patients will fill out an AUA symptom score questionnaire, have noninvasive uroflowmetry performed, and have a post-void residual measured by bladder scan. Using standard statistical analysis, we will see if there is a difference in symptoms, post-void residual, or maximum flow rate between baseline and 7 months post-op. We will continue the study to evaluate long-term efficacy, dropout rate, and complications. An FDA approved flexible dosing regimen will be allowed for the duration of the study.

ELIGIBILITY:
Patients will be selected by the investigator and sub-investigator's patient population, and physician referrals. All patients will meet the inclusion/ exclusion criteria.

Inclusion Criteria

1. Male ≥40 years of age
2. Clinical signs and symptoms of frequency and urgency, enlarged prostate and urodynamic study consistent with overactive bladder.
3. IPSS >12, with IPSS QoL > 3 at screening visit.
4. Ability and willingness to correctly complete the micturition diary and all the trial related questionnaires comply with scheduled visits and comply with trial procedures.
5. Capability of understanding and having signed the informed consent form after full discussion of the research, nature of the treatment, and its risks and benefits.
6. Procedure to treat BOO by TURP or PVP greater than or equal to 1 month ago.

Exclusion Criteria

1. A known history of interstitial cystitis, uninvestigated hematuria, or bladder outlet obstruction due to: mullerian duct cysts, urethral obstruction due to stricture/valves/sclerosis of urethral tumor, radiation cystitis, genitourinary tuberculosis, bladder calculi, or detrusor-sphincter dyssynergia.
2. Evidence of Urinary Tract Infection according to local standard of care.
3. Expectation of initiating treatment during the duration of this study with - any drug treatment for OAB, any drugs with significant anticholinergic, antispasmodic, parasympathetic, or cholinergic agonistic effects.
4. Use of any electrostimulation within the 30 days before randomization, or the expectation to initiate such therapy during the study.
5. Any condition which, in the opinion of the investigator, makes the patient unstable, or with contraindications for inclusion, e.g., uncontrolled narrow-angled glaucoma, urinary retention, preplanned prostate surgery, or gastric retention.
6. Significant hepatic or renal disease, defined as twice the upper limit of the reference ranges regarding serum concentrations of AST, ALT, ALP, urea nitrogen, or creatinine.
7. Use of any other investigational drug in the 2 months preceding visit 1.
8. History of postural hypotension or syncope in the judgement of the investigator based on local standards of care.
9. Alcohol and/or any other drug abuse in the opinion of the investigator.
10. Medications such as erythromycin, Biaxin (Clarithromycin), Sporanox (itraconazole), Nizoral (ketoconazole), Neoral and Sandimmune (cyclosporine), Velban (vinblastine) and miconazole.
11. Non-medication treatments such as bio-feedback or other bladder training exercises.

Ages: 40 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Te, MD, Principal Investigator — Cornell University
Locations (1):
- New York Hospital, Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Toviaz (Fesoterodine)
Started | 17
Completed | 11
Not Completed | 6
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Arm/Group | Toviaz (Fesoterodine)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 72.1 [53 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 17
BMI [Mean (Full Range); unit: kg/m^2] | 28.3 [19.1 to 35.9]
Voided Volume [Mean (Full Range); unit: mL] | 86 [20 to 292]
Laser [Number; unit: participants] | 13
TURP [Number; unit: participants] — Transurethral Resection of the Prostate
  participants | 4

OUTCOME MEASURES:

1. Primary Outcome: IPSS Obstructive
Description: International Prostate Symptom Score (IPSS) -is a 7 point scale used to screen, track and manage symptoms associated with BPH for obstructive, irritative, nocturia. The symptoms questions include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. Scores range from 1 to 5 for a total of maximum 35 points (0-7 Mildly symptomatic, 8-19 Moderately symptomatic, 20-35 Severely symptomatic). This measure was taken for patients with obstructive symptoms which includes hesitancy or difficulty initiating the stream, straining to void, a reduced flow, an intermittent stream or a sensation of incomplete emptying.
Time Frame: screening (Month 0), 2-months, 3-months, 7-months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IPSS Obstructive: Obstructive description
  Toviaz 4mg to 8mg
  Toviaz (Fesoterodine): 4mg to 8mg by mouth once daily
Arm/Group | IPSS Obstructive
Number analyzed (Participants) | 17
units on a scale
  Time Screening Month-0 | 9.1 (3.9)
  Time Month-2 | 7.5 (5.1)
  Time Month-3 | 8.4 (4.1)
  Time Month-7 | 7.9 (4.3)

2. Primary Outcome: IPSS Irritative
Description: International Prostate Symptom Score (IPSS) -is a 7 point scale used to screen, track and manage symptoms associated with BPH for obstructive, irritative, nocturia. The symptoms questions include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. Scores range from 1 to 5 for a total of maximum 35 points (0-7 Mildly symptomatic, 8-19 Moderately symptomatic, 20-35 Severely symptomatic). This measure was taken for patients with irritative symptoms which includes frequency, urgency, nocturia and urge incontinence
Time Frame: screening (Month 0), 2-months, 3-months, 7-months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IPSS Irritative: Irritative description
  Toviaz 4mg to 8mg
  Toviaz (Fesoterodine): 4mg to 8mg by mouth once daily
Arm/Group | IPSS Irritative
Number analyzed (Participants) | 17
units on a scale
  Time Screening Month-0 | 6.6 (2.1)
  Time Month-2 | 5.6 (2.6)
  Time Month-3 | 5.1 (2.2)
  Time Month-7 | 4.4 (2.4)

3. Primary Outcome: IPSS Nocturia
Description: International Prostate Symptom Score (IPSS) -is a 7 point scale used to screen, track and manage symptoms associated with BPH for obstructive, irritative, nocturia. The symptoms questions include feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. Scores range from 1 to 5 for a total of maximum 35 points (0-7 Mildly symptomatic, 8-19 Moderately symptomatic, 20-35 Severely symptomatic). This measure was taken for patients with nocturia meaning individuals who wake up during sleeping hours to urinate.
Time Frame: screening (Month 0), 2-months, 3-months, 7-months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IPSS Nocturia: Nocturia description
  Toviaz 4mg to 8mg
  Toviaz (Fesoterodine): 4mg to 8mg by mouth once daily
Arm/Group | IPSS Nocturia
Number analyzed (Participants) | 17
units on a scale
  Time Screening Month-0 | 3.2 (1.6)
  Time Month-2 | 2.8 (1.6)
  Time Month-3 | 2.6 (1.3)
  Time Month-7 | 2.6 (1.3)

4. Primary Outcome: International Prostate Symptom Score (IPSS) Quality of Life (QoL)
Description: IPSS Quality of Life (QoL) is one question used to assess how the patient's symptoms affect their quality of life. A score ranges from 1 to 6, with 6 being the worse outcome.
Time Frame: screening (Month 0), 2-months, 3-months, 7-months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IPSS QoL: QoL description
  Toviaz 4mg to 8mg
  Toviaz (Fesoterodine): 4mg to 8mg by mouth once daily
Arm/Group | IPSS QoL
Number analyzed (Participants) | 17
units on a scale
  Time Screening Month-0 | 4.2 (1.1)
  Time Month-2 | 3.8 (1.3)
  Time Month-3 | 3.5 (1.5)
  Time Month-7 | 3.5 (1.5)

5. Primary Outcome: Maximum Flow Rate (Qmax)
Description: Urodynamics was used to meause maximum flow rate (Qmax) which is the maximum recorded flow rate of urinary
Time Frame: screening (Month 0), 2-months, 3-months, 7-months
Measure: Mean (Standard Deviation); unit: mL/s
Groups:
- Qmax: Qmax
  Toviaz 4mg to 8mg
  Toviaz (Fesoterodine): 4mg to 8mg by mouth once daily
Arm/Group | Qmax
Number analyzed (Participants) | 17
mL/s
  Time Screening Month-0 | 15.3 (18.0)
  Time Month-2 | 10.2 (3.5)
  Time Month-3 | 10.6 (3.9)
  Time Month-7 | 10.5 (4.2)

6. Primary Outcome: Average Flow Rate (Qavg)
Description: Average (mean) flow rate (Qavg) is the the volume of urine voided divided by the continuous flow time
Time Frame: screening (Month 0), 2-months, 3-months, 7-months
Measure: Mean (Standard Deviation); unit: mL/s
Groups:
- QAvg: QAvg
  Toviaz 4mg to 8mg
  Toviaz (Fesoterodine): 4mg to 8mg by mouth once daily
Arm/Group | QAvg
Number analyzed (Participants) | 17
mL/s
  Time Screening Month-0 | NA (NA) — At the time that Qavg was collected, the Qavg data was skewed and was seen to be irrelevant and thus not reported for the screening appointment.
  Time Month-2 | 5.1 (2.0)
  Time Month-3 | 6.1 (2.6)
  Time Month-7 | 6.2 (3.0)

7. Primary Outcome: Postvoid Residual Volume (PVR)
Description: Postvoid residual volume (PVR) is the volume of fluid remaining in the bladder immediately after the completion of micturition.
Time Frame: screening (Month 0), 2-months, 3-months, 7-months
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Post-void Residual Volume (PVR): PVR
  Toviaz 4mg to 8mg
  Toviaz (Fesoterodine): 4mg to 8mg by mouth once daily
Arm/Group | Post-void Residual Volume (PVR)
Number analyzed (Participants) | 17
mL
  Time Screening Month-0 | 42.9 (43.2)
  Time Month-2 | 33.1 (39.4)
  Time Month-3 | 48.2 (64.8)
  Time Month-7 | 55.2 (56.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the study period which was 7-months.
Arm/Group | Toviaz (Fesoterodine)
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Toviaz (Fesoterodine) (N=17)
Constipation/Dry Mouth (Gastrointestinal disorders) | 3
Nausea/Vomiting (Gastrointestinal disorders) | 1
Urinary Leakage (Renal and urinary disorders) | 2

LIMITATIONS AND CAVEATS:
Small Sample size and the nonrandomized and nonblinded administration of the drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No